CLINICAL TRIAL: NCT02120014
Title: A Prospective Study to Determine the Association of Quantitated Blood and Plasma (Intravascular) Volume to Right Heart Hemodynamics, Venous Capacitance, and Regulatory Neurohormones in Patients With Chronic Heart Failure of Reduced and Preserved Ejection Fraction
Brief Title: Blood Volume and Hemodynamic Analysis in Patients With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Wayne L. Miller, M.D., Ph.D., Professor of Medicine, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13-003912
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Congestive Heart Failure
Keywords: Heart Failure; Heart Failure Reduced Ejection Fraction; Heart Failure Preserved Ejection Fraction; Venous Plethysmography; Blood Volume Study
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic; Heart Failure, Diastolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heart Failure Reduced EF (Experimental): Patient prior to clinically ordered right heart catheterization identified patients will have a blood volume measurement completed in the nuclear medicine laboratory. Patients will receive an intravenous administration of low dose iodinated I-131 labeled albumin. Blood specimens (6 cc each) will be drawn at 6 minute intervals times 6. The analysis will be completed following the testing.
  Venous plethysmography will be completed on eligible patients prior to the clinically indicated right heart catheterization. Calf and forearm venous compliance will be measured.
  Measurements form the right heart catheterization will be recorded for analysis.
  Interventions: Procedure: blood volume measurement; Procedure: venous plethysmography
- Heart Failure Preserved EF (Experimental): Patient prior to clinically ordered right heart catheterization identified patients will have a blood volume measurement completed in the nuclear medicine laboratory. Patients will receive an intravenous administration of low dose iodinated I-131 labeled albumin. Blood specimens (6 cc each) will be drawn at 6 minute intervals times 6. The analysis will be completed following the testing.
  Venous plethysmography will be completed on eligible patients prior to the clinically indicated right heart catheterization. Calf and forearm venous compliance will be measured.
  Measurements form the right heart catheterization will be recorded for analysis.
  Interventions: Procedure: blood volume measurement; Procedure: venous plethysmography

INTERVENTIONS:
Procedure: blood volume measurement — Patients will drink a solution 30 minutes prior to the test. They will need to lie still on a flat surface for 15 minutes. During the blood volume analysis portion of the test, a small amount of a radioactive isotope or tracer is injected.Blood samples are taken at 6 time points during the test. The blood volume test is used to measure the amount of blood in the patients body.
  A hematocrit measurement is done on the blood samples taken. This blood test calculates the percentage of red blood cells in the bloodstream.
  Other Names: Blood Volume - Red Cell Mass
Procedure: venous plethysmography — venous plethysmography is a non-invasive test to measure how well your veins and arteries in your forearm and calf work. Cuffs similar to blood pressure cuffs are placed on the upper and lower arm and the thigh and calf. Measurements are taken

SUMMARY:
The primary hypothesis is that patients with HFREF (heart failure with reduced ejection fraction) will demonstrate a markedly expanded intravascular volume which will correlate with elevated right heart hemodynamics and increased venous capacitance parameters, whereas patients with HFPEF(heart failure with preserved ejection fraction) will demonstrate euvolemia to mild volume expansion and a lack of correlation with hemodynamic and venous compliance parameters.

DETAILED DESCRIPTION:
The purpose of this study is to learn more about how the heart, blood vessels and blood volume interact in patients with heart failure and how measuring blood volume and vein capacity may help us develop better ways of treating and managing heart failure patients. This study will use two tests to measure blood volume and test the capacity of your veins and arteries in your limbs.

The blood volume test (also called a plasma volume test or a red cell mass test) is a standard clinical nuclear lab procedure used to measure the volume (amount) of blood in the body. The test also measures the volume of plasma and of red cells in the blood.

The other test is called a venous plethysmography, which is a non-invasive test to measure how well your veins and arteries in your forearm and calf work. Venous plethysmography measures the changes in the dimensions of your limbs by the use of strain gauges placed on the skin.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* patients identified with heart failure and diagnosed clinically to require right heart hemodynamic evaluation, New York Heart Association functional Class II-IV status/Stage C-D heart failure
* ischemic or nonischemic etiology heart failure
* left ventricular ejection fraction measured within 6 months of study enrollment

Exclusion Criteria:

* known significant intrinsic chronic kidney disease (baseline Glomerular Filtration Rate <15 ml/min/1.73m²) or patients receiving hemodialysis
* known renal artery stenotic disease
* females who are pregnant
* allergy to iodine contrast, intravenous pyelogram dye, shellfish or eggs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-04-21 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Total Blood Volume Measurement | Baseline prior to a clinically indicated right heart catheterization.
  Blood volume will be measured at baseline for eligible patients prior to a clinical right heart catheterization.

SECONDARY OUTCOMES:
venous plethysmography | Baseline prior to a clinically indicated right heart catheterization.
  venous plethysmography will be measured at baseline for eligible patients prior to a clinical right heart catheterization.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne L Miller, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States